CLINICAL TRIAL: NCT00757471
Title: Membranepeeling With Brillant Blue Versus Membranepeeling With Indocyanine Green for Patients With Idiopathic Macular Holes.
Brief Title: Brillant Blue Versus Indocyanine Green for Macular Hole Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Principal Investigator, Dr. Christiane I. Falkner-Radler, MD, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR-5-CI-2008
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Idiopathic Macular Holes
Keywords: Macular hole surgery; membranepeeling; closure rate; vitreoretinal dyes
MeSH Terms: interventions — procion brilliant blue HGR; Indocyanine Green

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Brillant Blue
  Interventions: Procedure: Brillant Blue
- Group 2 (Active Comparator): Indocyanine Green
  Interventions: Procedure: Indocyanine Green

INTERVENTIONS:
Procedure: Brillant Blue — Membrane Peeling with Brillant Blue
  Arms: Group 1
Procedure: Indocyanine Green — Membrane Peeling with indocyanine Green
  Arms: Group 2

SUMMARY:
Macular Hole Surgery with two different Dyes

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic stage 3 and 4 macular holes
* Stage 2 macular holes, followed up for at least 6 months
* Pseudophakic and phakic eyes
* Age over 60 years

Exclusion Criteria:

* Traumatic macular holes
* Secondary macular holes
* Severe ocular diseases

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Macular Hole Closure Rate | 12 Months

SECONDARY OUTCOMES:
Visual Acuity Microperimetry Optical Coherence Tomography | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kreppler, MD, Study Chair — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery; Christiane I Falkner-Radler, MD, Principal Investigator — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Locations (1):
- The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser surgery, Vienna, Vienna, Austria